CLINICAL TRIAL: NCT04910217
Title: Robot-Assisted Gait Therapy in the Subacute Phase of First Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Collaborators: Masaryk University (Other); VSB - Technical University of Ostrava (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-Lokowalkers-2021
Record Dates: First submitted 2021-05-20; First posted 2021-06-02 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Ischemic Stroke
Keywords: gait; stroke; robotic rehabilitation; exoskeleton; neurorehabilitation; Lokomat
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: Single-centre randomized parallel group neurorehabilitation trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lokomat intervention (Experimental): Patients randomized into the Lokomat arm will undergo therapy with Lokomat Pro FreeD for 20-50 minutes 5-times a week, a total of 15-times during the in-hospital stay in a total time of 1,800 minutes.
  Interventions: Procedure: Conventional rehabilitation; Procedure: Lokomat intervention
- Conventional rehabilitation (Experimental): Patients in this arm will undergo conventional rehabilitation ((ergotherapy and physiotherapy) for 60 min 5 times a week, a total of 15 times within 3 weeks (a total of 1200 min)
  Interventions: Procedure: Conventional rehabilitation; Procedure: Leg/lower body exerciser device intervention.

INTERVENTIONS:
Procedure: Conventional rehabilitation — Patients will undergo conventional rehabilitation
Procedure: Leg/lower body exerciser device intervention. — Patients will undergo leg/lower body exerciser device therapy.
  Arms: Conventional rehabilitation
Procedure: Lokomat intervention — Patients will undergo therapy with Lokomat Pro FreeD device intervention.
  Arms: Lokomat intervention

SUMMARY:
Robot-assisted gait training (RAGT) represents a modern concept of neurorehabilitation in stroke patients. This single-center randomized parallel-group neurorehabilitation trial with blinded primary outcome assessment is aimed at patients after the first-ever ischaemic stroke in the anterior or posterior cerebral circulation.

DETAILED DESCRIPTION:
The main aim is to determine, whether the RAGT by using the Lokomat exoskeleton device (Hoccoma, Switzerland) plus the protocol-defined conventional rehabilitation versus conventional rehabilitation improves the gait of post-stroke patients after 6 months. Both groups are treated with the protocol-defined rehabilitation (ergotherapy and physiotherapy) for 60 min 5 times a week, a total of 15 times within 3 weeks (a total of 1200 min). The Lokowalkers group undergoes the RAGT using the Lokomat Pro Freed device for 20-50 minutes 5 times a week for a total of 15 times for 3 weeks (a total of 1800 minutes). The primary endpoint is the Functional Ambulation Category (FAC) after 3 months. Secondary endpoints include FAC (after 15th therapy), 10-meter walk test (10MWT) (after 15th therapy, after 3 months), Timed Up and Go Test (TUG) (after 15th therapy and after 3 months, 3-months modified Rankin Scale (mRS), and Berg Balance Scale (BBS, after 15th therapy, after 3 months).

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent by the participant or legal representative
* interval between stroke and first rehabilitation session < 6 weeks (study target within 2 weeks)
* age > 18 years
* early modified Rankin scale (mRS) 2 to 4 (pre-stroke mRS 0 to 1)
* early FAC of 0 to 3 (pre-stroke FAC of 5)
* standing ability with support up to 3 minutes and vertical tolerance > 15 minutes

Exclusion Criteria:

* inability or refusal to sign an informed consent
* history of stroke or another brain disease (tumour, multiple sclerosis, brain or spinal cord injury)
* severe internal, oncological, or surgical comorbidity preventing long-term re-habilitation or causing chronic or progressive gait disorder
* limited collaboration of any reason, moderate or severe dementia assessed by using the Montreal Cognitive Assessment (MoCA) scale
* impaired skin integrity in the lower torso and limbs preventing the use of Lokomat device
* limitations given by the Lokomat exoskeleton device (weight > 135 kg, thigh-length 23-35 cm, shank length 35-47cm)
* limitations given by the leg/lower body exerciser (weight > 180 kg, height < 120 cm or > 200 cm, (sub)acute lower limb fractures, deep vein thrombosis, skin disintegration)
* any contraindication to perform brain MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Functional Ambulation Category (FAC) at 3 months | 3 months
  Functional Ambulation Category (FAC) - the scale range is from 0 to 5. The value at 6-months will be observed.

SECONDARY OUTCOMES:
Functional Ambulation Category (FAC) (after 3 weeks) | 3 weeks
  Functional Ambulation Category (FAC) - the scale range is from 0 to 5. The value after 3 weeks will be observed.
10-meter walk test (10-MWT) (after 3 weeks and 3 months) | up to 3 months
  10-meter walk test will be performed after 3 weeks and 3 months
Timed Up and Go Test (TUG) (after 3 weeks, after 3 months) | up to 3 months
  Timed Up and Go Test (TUG) will be performed after 3 weeks, after 3 months
3-months modified Rankin Scale (mRS) | up to 3 months
  3-months modified Rankin Scale (mRS) assesses the functional independence and represents a standard outcome measure in post-stroke patients (range from 0 to 6).
Berg Balance Scale (BBS, after 3 weeks, after 3 months) | up to 3 months
  Berg Balance Scale (BBS) objectifies balance functions in 14 tasks. It assesses the risk of possible falls: 0-20 high, 21-40 medium, 41-56 low risk of falling.
Adverse effects | up to 3 years
  The number and character of adverse effects will be observed during the study.
Early termination of the study | up to 3 years
  The number of patients terminating the study early will be observed during the study.
Reason/s for the termination | up to 3 years
  The reason/s for the termination will be observed during the study.
Study-related death or death unrelated to study | up to 3 years
  The number of study-related deaths or deaths unrelated to study will be observed during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ondřej Volný, MD,PhD,FESO, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehrholz J, Wagner K, Rutte K, Meissner D, Pohl M. Predictive validity and responsiveness of the functional ambulation category in hemiparetic patients after stroke. Arch Phys Med Rehabil. 2007 Oct;88(10):1314-9. doi: 10.1016/j.apmr.2007.06.764. PMID 17908575
- [Background] Albert SJ, Kesselring J. Neurorehabilitation of stroke. J Neurol. 2012 May;259(5):817-32. doi: 10.1007/s00415-011-6247-y. Epub 2011 Oct 1. PMID 21964750
- [Background] Winstein CJ, Stein J, Arena R, Bates B, Cherney LR, Cramer SC, Deruyter F, Eng JJ, Fisher B, Harvey RL, Lang CE, MacKay-Lyons M, Ottenbacher KJ, Pugh S, Reeves MJ, Richards LG, Stiers W, Zorowitz RD; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Jun;47(6):e98-e169. doi: 10.1161/STR.0000000000000098. Epub 2016 May 4. PMID 27145936
- [Background] Maier M, Ballester BR, Verschure PFMJ. Principles of Neurorehabilitation After Stroke Based on Motor Learning and Brain Plasticity Mechanisms. Front Syst Neurosci. 2019 Dec 17;13:74. doi: 10.3389/fnsys.2019.00074. eCollection 2019. PMID 31920570
- [Background] Morone G, Paolucci S, Cherubini A, De Angelis D, Venturiero V, Coiro P, Iosa M. Robot-assisted gait training for stroke patients: current state of the art and perspectives of robotics. Neuropsychiatr Dis Treat. 2017 May 15;13:1303-1311. doi: 10.2147/NDT.S114102. eCollection 2017. PMID 28553117
- [Background] Moucheboeuf G, Griffier R, Gasq D, Glize B, Bouyer L, Dehail P, Cassoudesalle H. Effects of robotic gait training after stroke: A meta-analysis. Ann Phys Rehabil Med. 2020 Nov;63(6):518-534. doi: 10.1016/j.rehab.2020.02.008. Epub 2020 Mar 27. PMID 32229177
- [Background] Jorgensen HS, Nakayama H, Raaschou HO, Olsen TS. Recovery of walking function in stroke patients: the Copenhagen Stroke Study. Arch Phys Med Rehabil. 1995 Jan;76(1):27-32. doi: 10.1016/s0003-9993(95)80038-7. PMID 7811170
- [Background] Bruni MF, Melegari C, De Cola MC, Bramanti A, Bramanti P, Calabro RS. What does best evidence tell us about robotic gait rehabilitation in stroke patients: A systematic review and meta-analysis. J Clin Neurosci. 2018 Feb;48:11-17. doi: 10.1016/j.jocn.2017.10.048. Epub 2017 Dec 6. PMID 29208476
- [Background] Kim MS, Kim SH, Noh SE, Bang HJ, Lee KM. Robotic-Assisted Shoulder Rehabilitation Therapy Effectively Improved Poststroke Hemiplegic Shoulder Pain: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2019 Jun;100(6):1015-1022. doi: 10.1016/j.apmr.2019.02.003. Epub 2019 Mar 13. PMID 30878496
- [Background] Mehrholz J, Thomas S, Kugler J, Pohl M, Elsner B. Electromechanical-assisted training for walking after stroke. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD006185. doi: 10.1002/14651858.CD006185.pub5. PMID 33091160
- [Background] Zaidi SF, Aghaebrahim A, Urra X, Jumaa MA, Jankowitz B, Hammer M, Nogueira R, Horowitz M, Reddy V, Jovin TG. Final infarct volume is a stronger predictor of outcome than recanalization in patients with proximal middle cerebral artery occlusion treated with endovascular therapy. Stroke. 2012 Dec;43(12):3238-44. doi: 10.1161/STROKEAHA.112.671594. Epub 2012 Nov 15. PMID 23160876
- [Background] Bucker A, Boers AM, Bot JCJ, Berkhemer OA, Lingsma HF, Yoo AJ, van Zwam WH, van Oostenbrugge RJ, van der Lugt A, Dippel DWJ, Roos YBWEM, Majoie CBLM, Marquering HA; MR CLEAN Trial Investigators (Multicenter Randomized Clinical Trial of Endovascular Treatment for Acute Ischemic Stroke in the Netherlands). Associations of Ischemic Lesion Volume With Functional Outcome in Patients With Acute Ischemic Stroke: 24-Hour Versus 1-Week Imaging. Stroke. 2017 May;48(5):1233-1240. doi: 10.1161/STROKEAHA.116.015156. Epub 2017 Mar 28. PMID 28351963
- [Background] Aurich-Schuler T, Gut A, Labruyere R. The FreeD module for the Lokomat facilitates a physiological movement pattern in healthy people - a proof of concept study. J Neuroeng Rehabil. 2019 Feb 6;16(1):26. doi: 10.1186/s12984-019-0496-x. PMID 30728040
- [Background] Bower K, Thilarajah S, Pua YH, Williams G, Tan D, Mentiplay B, Denehy L, Clark R. Dynamic balance and instrumented gait variables are independent predictors of falls following stroke. J Neuroeng Rehabil. 2019 Jan 7;16(1):3. doi: 10.1186/s12984-018-0478-4. PMID 30612584
- [Background] Heinemann AW, Linacre JM, Wright BD, Hamilton BB, Granger C. Relationships between impairment and physical disability as measured by the functional independence measure. Arch Phys Med Rehabil. 1993 Jun;74(6):566-73. doi: 10.1016/0003-9993(93)90153-2. PMID 8503745
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055
- [Background] Anderson C, Laubscher S, Burns R. Validation of the Short Form 36 (SF-36) health survey questionnaire among stroke patients. Stroke. 1996 Oct;27(10):1812-6. doi: 10.1161/01.str.27.10.1812. PMID 8841336
- [Background] Park IJ, Park JH, Seong HY, You JSH, Kim SJ, Min JH, Ko HY, Shin YI. Comparative Effects of Different Assistance Force During Robot-Assisted Gait Training on Locomotor Functions in Patients With Subacute Stroke: An Assessor-Blind, Randomized Controlled Trial. Am J Phys Med Rehabil. 2019 Jan;98(1):58-64. doi: 10.1097/PHM.0000000000001027. PMID 30142092
- [Background] Barca C, Foray C, Hermann S, Doring C, Schafers M, Jacobs AH, Zinnhardt B. Characterization of the inflammatory post-ischemic tissue by full volumetric analysis of a multimodal imaging dataset. Neuroimage. 2020 Nov 15;222:117217. doi: 10.1016/j.neuroimage.2020.117217. Epub 2020 Jul 31. PMID 32745676
- [Background] Baudat C, Marechal B, Corredor-Jerez R, Kober T, Meuli R, Hagmann P, Michel P, Maeder P, Dunet V. Automated MRI-based volumetry of basal ganglia and thalamus at the chronic phase of cortical stroke. Neuroradiology. 2020 Nov;62(11):1371-1380. doi: 10.1007/s00234-020-02477-x. Epub 2020 Jun 17. PMID 32556424
- [Background] Bernarding J, Braun J, Hohmann J, Mansmann U, Hoehn-Berlage M, Stapf C, Wolf KJ, Tolxdorff T. Histogram-based characterization of healthy and ischemic brain tissues using multiparametric MR imaging including apparent diffusion coefficient maps and relaxometry. Magn Reson Med. 2000 Jan;43(1):52-61. doi: 10.1002/(sici)1522-2594(200001)43:13.0.co;2-5. PMID 10642731
- [Derived] Fiedorova I, Banikova S, Adamec T, Konde A, Hanzlikova P, Ganesh A, Bar M, Volny O. Robot-Assisted Gait Therapy in the Subacute Phase of Ischemic Stroke: A Randomized Controlled Trial. Ann Indian Acad Neurol. 2025 Nov 28. doi: 10.4103/aian.aian_526_25. Online ahead of print. PMID 41313041